CLINICAL TRIAL: NCT04042272
Title: Evaluation of s100β, NSE and Glial Fibrillary Acidic Protein Levels in Preoperative and Postoperative Renal Transplantation
Brief Title: Evaluation of s100β, NSE and GFAP Levels in Renal Transplantation
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Bora Dinc, Assistant Professor Department of Anesthesiology and Reanimation, Akdeniz University
Other Study IDs: S100β, NSE n GFAP in RT
Record Dates: First submitted 2019-07-31; First posted 2019-08-01 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Kidney Transplant; Complications; Neurologic Manifestations; Uremic Encephalopathy
Keywords: kidney transplantation; s100β; neuron specific enolase; glial fibrillary acidic protein
MeSH Terms: conditions — Neurologic Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — s100β, neuron specific enolase and glial fibrillary acidic
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy volunteers: Healthy volunteers group; Kidney donor groups; Course of the research: Blood samples from all groups shall be taken for S100β, NSE, and GFAP in the preoperative period, in the operating room and after 1st, 7th day and the first following month in the postoperative period. Mortality and morbidity of the patients shall be recorded. Neurological damage and its effect on prognosis shall be examined within the patients with S100β, NSE, and GFAP. Patients' demographic data, accompanying diseases, American Society of Anesthesiology classification, main etiology, preoperative laboratory values shall be recorded accordingly. In addition, routinely taken anesthetics, duration of the operation, duration of anesthesia, duration before the reperfusion, duration of postperfusion, graft hot and cold ischemia durations, first measured central venous pressure, volume replacement therapy, blood component transfusion, and immunosuppressive drugs are given during the operation shall be recorded.
  Interventions: Diagnostic Test: S100β, Neuron specific enolase (NSE) and Glial fibrillary acidic protein (GFAP)
- Living kidney graft recipients: Kidney transplant group; Course of the research: Course of the research: Blood samples from all groups shall be taken for S100β, NSE, and GFAP in the preoperative period, in the operating room and after 1st, 7th day and the first following month in the postoperative period. Mortality and morbidity of the patients shall be recorded. Neurological damage and its effect on prognosis shall be examined within the patients with S100β, NSE, and GFAP. Patients' demographic data, accompanying diseases, American Society of Anesthesiology classification, main etiology, preoperative laboratory values shall be recorded accordingly. In addition, routinely taken anesthetics, duration of the operation, duration of anesthesia, duration before the reperfusion, duration of postperfusion, graft hot and cold ischemia durations, first measured central venous pressure, volume replacement therapy, blood component transfusion, and immunosuppressive drugs are given during the operation shall be recorded.
  Interventions: Diagnostic Test: S100β, Neuron specific enolase (NSE) and Glial fibrillary acidic protein (GFAP)

INTERVENTIONS:
Diagnostic Test: S100β, Neuron specific enolase (NSE) and Glial fibrillary acidic protein (GFAP) — S100β is 10.4 kDa protein. Synthesized with end-feet processes of astrocytes in the brain S100β belongs to low molecular weight EF-hand type acidic calcium-binding protein superfamily. This protein is metabolized in the kidneys and removed with urine. It is shown that S100β does not show differences due to ethnical groups or genders and is not affected by circadian rhythm. Although S100β is also found in other tissues, it is in higher concentrations in the brain so it can be used as an early indicator for brain damage.NSE is an SSS protein which exists in neurons and neuroendocrine tissues. NSE plays a role in glycolytic route in neurons as intracytoplasmic enzyme increasing serum level in case of neuron damage. Whilst S100β is the marker of astroglia dysfunction, NSE is the marker of neuronal dysfunction. Glial fibrillary acidic protein (GFAP) is the intermediate filament cell skeleton protein found in astrocytes. It originates from the same root structure as S100β.

SUMMARY:
Uremic encephalopathy is an organic brain disorder may be frequently seen in patients with acute or chronic renal failure. Certain neurological symptoms can be found under clinical glomerular filtration rate of 15 ml/minutes. The above mentioned neurological disorders can be due to uremic toxins as well as many other reasons such as metabolic and hemodynamic disturbances, inflammation, or oxidative stress. Most frequent symptoms are impaired consciousness, lethargy, cranial nerve involvement, nystagmus, dysarthria, and even coma and death. Brain tissue may receive damage and some secondary biomarkers may appear in case BUN (Blood Urea Nitrogen) level is >175 mg/dl together with neuroinflammation. Although hemodialysis is a temporary solution in terms of treatment, these symptoms may be reversible in the long-run with organ transplantation. A rigorous neurological assessment before transplantation is important for identifying the severity and distribution of the neurological disorder as well as defining the abnormalities that are responding to the current treatments and foreseeing potential postoperative prognosis.

S100β is excreted by astrocytes in brain damage cases. S100β level rises when brain damage starts, thus it may be used in the prognosis of brain damage in its early period. Neuron-specific enolase (NSE) functions as intracytoplasmic enzyme and serum level rises in neuron damage. Glial fibrillary acidic protein (GFAP), on the other hand, is the intermediary filament cytoskeleton protein found in astrocytes. It has the same root structure with S100β.

The purpose of this study is to assess neurological damage by looking at the levels of S100β, NSE and GFAP in patients who underwent kidney transplantation and to analyze the impacts on the prognosis.

DETAILED DESCRIPTION:
Encephalopathy, thiamine deficiency, uremia, hypertension, electrolyte imbalance after dialysis are clinical pictures with high incidences in case of renal failure. There are multifactor reasons in its pathophysiology such as hormonal imbalance, oxidative stress, accumulation of metabolites in time, disorders in excitatory and inhibitory transmitters and intermediary metabolisms.

Neurological disorders that affect renal transplant patients during the waiting list period do not only significantly affect preoperative morbidity and even mortality, but also show important predictive factors for neurological symptoms after the transplantation. A rigorous neurological assessment before transplantation is important for identifying the severity and distribution of the neurological disorder as well as defining the abnormalities that are responding to the current treatments and foreseeing potential postoperative prognosis. Specific indexes preferred for neurological assessment before the transplant may vary depending on the clinic; however, correct and differential diagnosis of various symptoms may be difficult despite the use of various diagnostic tools such as biochemical, neurophysiologic, neuropsychological and neuroimaging tools.

S100β is a 10.4 kDa protein. S100β is synthesized in the brain through endfeet processes of astrocytes and it belongs to the superfamily of low molecular weight EF-hand type acidic calcium-binding proteins. This protein is metabolized in the kidneys first and foremost and then discharged through urine. It has been shown that S100β does not differ depending on ethnic groups and genders and is not affected by circadian rhythm. Even though S100β may be found in other tissues, it may be used as an early marker for brain damage since it is found in higher concentration in the brain.

Astrocytes are the key agents for homeostasis regulation in the central nervous system (CNS) and they secrete S100β after brain damage. Certain studies show that increased levels of S100β may be used as an early marker of intracerebral changes in the brains of patients with acute or chronic liver failure and hepatic encephalopathy (HE) before the development of cerebral edema.

Moreover, some studies suggest that increased levels of S100β in serum concentrations may predict HE. However, there are few pieces of evidence that prove the correlation between S100β levels and HE's presence.

NSE (neuron-specific enolase) is a CNS protein found in neurons and neuroendocrine tissues. NSE functions in the glycolytic path of neurons as an intracytoplasmic enzyme and its serum levels increase in case of neuron damage. S100β is a marker of astroglial dysfunction while NSE is a marker of neuronal dysfunction.

And Glial fibrillary acidic protein (GFAP) is reported to be more specific to brain tissue compared to S100β. There are studies showing that prognosis is worse when both GFAP and S100β levels are seen to increase in the assessment of neurological damage, especially in cases of head traumas, thus supporting the use of both proteins for higher prognostic accuracy. GFAP is also a biomarker used for neurodegenerative diseases and ischemic cases other than cases of trauma.

The aim of the present study is to analyze neurological damage in renal transplant patients through S100β, NSE and GFAP serum concentrations and assess their impacts on the prognosis.

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal failure patients
* Healthy volunteer patients.

Exclusion Criteria:

* Nonvolunteers
* Active infections
* Oncologic or hematologic diseases
* Cadaver graft recipients
* History with psychoactive medications
* History with a respiratory system or central nervous system disorders
* Severe heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients' demographic data (age, gender, weight, height), accompanying diseases, ASA classification, main etiology, preoperative serums taken in the preoperative period; serum sodium, potassium, ammonium, total bilirubin, ALT, AST, albumin, alkaline phosphatase, INR, creatinine, and BUN shall be recorded accordingly. In addition, routinely taken anesthetics, duration of the operation, duration of anesthesia, duration before the reperfusion, duration of postperfusion, graft hot and cold ischemia durations, first measured central venous pressure, volume replacement therapy, blood component transfusion, total fluid amount given during the operation, corticosteroids and immunosuppressive drugs given during the operation shall be recorded.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Assessment of serum s100β | 2 years
  Approximately 40 patients planned to have living donor renal transplantation and 40 patients planned to have nephrectomy for kidney donation will be included in the study.
  The blood samples are taken in the preoperative period before the induction of anesthesia in the operating room and postoperative (the first day, the seventh day and the first month) period to analyze S100β serum concentrations and neurologic damage of kidney transplantation and nephrectomy patients besides evaluating its effect on prognosis. These samples shall be kept at -80 0C until plasma separation process.
Assessment of serum NSE | 2 years
  Approximately 40 patients planned to have living donor renal transplantation and 40 patients planned to have nephrectomy for kidney donation will be included in the study.
  The blood samples are taken in the preoperative period before the induction of anesthesia in the operating room and postoperative (the first day, the seventh day and the first month) period to analyze NSE serum concentrations and neurologic damage of kidney transplantation and nephrectomy patients besides evaluating its effect on prognosis. These samples shall be kept at -80 0C until plasma separation process.
Assessment of serum GFAP | 2 years
  Approximately 40 patients planned to have living donor renal transplantation and 40 patients planned to have nephrectomy for kidney donation will be included in the study.
  The blood samples are taken in the preoperative period before the induction of anesthesia in the operating room and postoperative (the first day, the seventh day and the first month) period to analyze GFAP serum concentrations and neurologic damage of kidney transplantation and nephrectomy patients besides evaluating its effect on prognosis. These samples shall be kept at -80 0C until plasma separation process.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University Hospital, Antalya, Turkey (Türkiye)